CLINICAL TRIAL: NCT01531361
Title: A Phase I Trial of Sorafenib (CRAF, BRAF, KIT, RET, VEGFR, PDGFR Inhibitor) or Crizotinib (MET, ALK, ROS1 Inhibitor) in Combination With Vemurafenib (BRAF Inhibitor) in Patients With Advanced Malignancies
Brief Title: Vemurafenib With Sorafenib Tosylate or Crizotinib in Treating Patients With Advanced Malignancies With BRAF Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1183; NCI-2012-00217 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-1183 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-02-06; First posted 2012-02-10 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Advanced Malignant Neoplasm; BRAF Gene Mutation; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm; Refractory Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Neoplasms | interventions — Crizotinib; Sorafenib; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (vemurafenib and sorafenib tosylate) (Experimental): Patients receive vemurafenib PO BID and sorafenib tosylate PO BID on days 1-28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sorafenib Tosylate; Drug: Vemurafenib
- Arm II (vemurafenib and crizotinib) (Experimental): Patients receive vemurafenib as in Arm I and crizotinib PO QD or BID on days 1-28.
  Interventions: Drug: Crizotinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vemurafenib

INTERVENTIONS:
Drug: Crizotinib — Given PO
  Other Names: MET Tyrosine Kinase Inhibitor PF-02341066; PF-02341066; PF-2341066; Xalkori
  Arms: Arm II (vemurafenib and crizotinib)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Arm I (vemurafenib and sorafenib tosylate)
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX-4032; PLX4032; RG 7204; RG7204; RO 5185426; Zelboraf

SUMMARY:
This phase I clinical trial studies vemurafenib with sorafenib tosylate or crizotinib in treating patients with advanced malignancies with BRAF mutations. Sorafenib tosylate and crizotinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Sorafenib tosylate may also stop the growth of advanced malignancies by blocking blood flow to tumors. Drugs used in chemotherapy, such as vemurafenib, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving vemurafenib together with sorafenib tosylate or crizotinib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of sorafenib tosylate (sorafenib) or crizotinib in combination with vemurafenib in patients with advanced cancers who progressed on standard therapy.

SECONDARY OBJECTIVES:

I. Preliminary assessment of antitumor efficacy of sorafenib or crizotinib combination with vemurafenib in patients with advanced cancers.

II. Preliminary assessment of the pharmacokinetic (PK) profile of sorafenib or crizotinib in combination with vemurafenib.

III. Preliminary assessment of biomarkers.

OUTLINE: This is a dose-escalation study of vemurafenib and sorafenib tosylate. Patients are assigned to 1 of 2 treatment arms by their physician.

ARM I: Patients receive vemurafenib orally (PO) twice daily (BID) and sorafenib tosylate PO BID on days 1-28.

ARM II: Patients receive vemurafenib as in Arm I and crizotinib PO once daily (QD) or BID on days 1-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic cancers and BRAF mutations that are refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months; patients with BRAF mutation in cell free deoxyribonucleic acid (DNA) (tested in Clinical Laboratory Improvement Amendments [CLIA] lab) are also eligible
* Patients must be >= 3 weeks beyond treatment with a cytotoxic chemotherapy regimen, or therapeutic radiation, or major surgery; patients may have received palliative localized radiation immediately before or during treatment provided that radiation is not delivered to the only site of disease being treated under this protocol; for biologic/targeted agents patients must be >= 5 half-lives or >= 3 weeks from the last dose (whichever comes first); patients previously treated with vemurafenib monotherapy do not have to stop medication before they start on the protocol
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1,000/mL
* Platelets >= 75,000/mL
* Creatinine =< 2 X upper limit of normal (ULN)
* Total bilirubin =< 2 X ULN (exceptions may apply to benign non-malignant indirect hyperbilirubinemia such as Gilbert syndrome)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) and/or aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 5 X ULN
* Exception for patients with liver metastasis: total bilirubin =< 3 x ULN; ALT (SGPT) =< 8 X ULN
* Dermatology evaluation with excision of any suspicious lesions prior to initiation of therapy
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose
* Women of childbearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to initiation of therapy
* Life expectancy > 12 weeks in the opinion of the investigator
* Patients must be able to understand and be willing to sign a written informed consent document
* Patient must be able to swallow pills

Exclusion Criteria:

* Uncontrolled intercurrent illness, including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, need for ventilatory support
* Syndrome of congenital corrected QT interval (QTc) prolongation or QTc > 500 msec
* Patients with clinically significant cardiovascular disease: history of cerebrovascular accident (CVA) within 6 months, myocardial infarction or unstable angina within 6 months, or unstable angina pectoris
* Pregnant or lactating women
* History of hypersensitivity to vemurafenib
* History of hypersensitivity to sorafenib for vemurafenib/sorafenib arm
* History of hypersensitivity to crizotinib for vemurafenib/crizotinib arm
* History of hypersensitivity to any component of the formulation
* Patients unwilling or unable to sign informed consent document
* Patients using any of the following medications: mesoridazine, dronedarone, thioridazine, ziprasidone, levomethadyl, and saquinavir for vemurafenib/sorafenib arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vemurafenib and sorafenib tosylate or crizotinib, defined as the highest dose studied in which the incidence of dose limiting toxicity was less than 33% | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org